CLINICAL TRIAL: NCT00246350
Title: Dose-Response of Manipulation for Chronic Headache
Brief Title: Spinal Manipulation for Treatment of Chronic Headaches
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Western States (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT002324 (NIH); R21AT002324 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-10-31 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-11

CONDITIONS: Headache Disorders
Keywords: Headaches; Spinal manipulation; Massage; chiropractic
MeSH Terms: conditions — Headache Disorders; Headache | interventions — Massage; Manipulation, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): 8 light massage treatments
  Interventions: Procedure: massage
- 2 (Active Comparator): 16 light massage treatments
  Interventions: Procedure: massage
- 3 (Experimental): 8 spinal manipulation treatments
  Interventions: Procedure: spinal manipulation
- 4 (Experimental): 16 spinal manipulation treatments
  Interventions: Procedure: Spinal manipulation

INTERVENTIONS:
Procedure: massage — 8 light massage treatments and hot pack
  Arms: 1
Procedure: massage — 16 light massage treatments and hot packs
  Arms: 2
Procedure: spinal manipulation — 8 high velocity, low amplitude spinal manipulation treatments and hot pack
  Arms: 3
Procedure: Spinal manipulation — 16 high velocity, low amplitude spinal manipulation treatments and hot pack
  Arms: 4

SUMMARY:
This study will determine the effectiveness of spinal manipulation in reducing pain in people with chronic headaches accompanied by neck pain. This study will also determine the number of spinal manipulation treatments necessary for optimal pain relief.

DETAILED DESCRIPTION:
Spinal manipulation is the signature therapy of chiropractic care involving manual adjustment of joints in the neck and back. Data indicate that spinal manipulation is an effective treatment for back pain and chronic headaches, particularly cervicogenic headaches, which are caused by problems in the cervical spine. However, studies that have determined the optimal frequency and duration of spinal manipulation treatment are limited. This study will determine the feasibility of conducting a large spinal manipulation clinical trial. This study will also determine the effectiveness of spinal manipulation in treating cervicogenic headaches and neck pain and the optimal number of treatments necessary to sustain spinal manipulation benefits.

Participants will be randomly assigned to receive weekly sessions of either spinal manipulation or light massage treatments for 8 to 16 weeks. Self-report scales will be used to assess participants' headache frequency, pain, satisfaction with treatment, and overall physical and mental health. Assessments will occur at study entry, at the end of each week, and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* History of cervicogenic headaches

Exclusion Criteria:

* Contraindications to spinal manipulation or massage
* Use of chiropractic or therapeutic massage care prior to study entry
* Use of any prophylactic prescription medication
* Involved in any type of lawsuit prior to study entry
* Headaches with several different causes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Modified Von Korff pain scale for headaches

SECONDARY OUTCOMES:
Modified Von Korff disability scale for headaches
Number of cervicogenic headaches
general physical and mental health status
patient satisfaction
neck pain

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Haas, DC, Principal Investigator — University of Western States
Locations (1):
- Western States Chiropractic College, Portland, Oregon, United States

REFERENCES:
- [Background] Haas M, Groupp E, Aickin M, Fairweather A, Ganger B, Attwood M, Cummins C, Baffes L. Dose response for chiropractic care of chronic cervicogenic headache and associated neck pain: a randomized pilot study. J Manipulative Physiol Ther. 2004 Nov-Dec;27(9):547-53. doi: 10.1016/j.jmpt.2004.10.007. PMID 15614241
- [Result] Haas M, Spegman A, Peterson D, Aickin M, Vavrek D. Dose response and efficacy of spinal manipulation for chronic cervicogenic headache: a pilot randomized controlled trial. Spine J. 2010 Feb;10(2):117-28. doi: 10.1016/j.spinee.2009.09.002. PMID 19837005
- [Result] Haas M, Aickin M, Vavrek D. A preliminary path analysis of expectancy and patient-provider encounter in an open-label randomized controlled trial of spinal manipulation for cervicogenic headache. J Manipulative Physiol Ther. 2010 Jan;33(1):5-13. doi: 10.1016/j.jmpt.2009.11.007. PMID 20114095
- [Result] Haas M, Schneider M, Vavrek D. Illustrating risk difference and number needed to treat from a randomized controlled trial of spinal manipulation for cervicogenic headache. Chiropr Osteopat. 2010 May 24;18:9. doi: 10.1186/1746-1340-18-9. PMID 20497573
- [Result] Vavrek D, Haas M, Peterson D. Physical examination and self-reported pain outcomes from a randomized trial on chronic cervicogenic headache. J Manipulative Physiol Ther. 2010 Jun;33(5):338-48. doi: 10.1016/j.jmpt.2010.05.004. PMID 20605552